CLINICAL TRIAL: NCT04603456
Title: MicroRNA-155 Assay in Childhood Allergic Rhinitis Before and After Combined Sublingual Immunotherapy and Probiotics
Brief Title: miRNA-155 Assay Before and After Immunotherapy and Probiotics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Fedaa Nabil, Assisstant lecturer, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: miR-155 in allergic rhinitis
Record Dates: First submitted 2020-10-11; First posted 2020-10-26 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Intervention Model Description: Group I included 15 cases who received probiotics only. Group II included 15 children who received SLIT. Group III included 15 children who received probiotics and SLIT.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Probiotic Group (Experimental): consisted of 15 cases who received probiotics only. A drug called Lacteol fort (Rameda Company) . A sachet was taken once daily for three months. Each sachet contains 10 billions lactobacilli.
  Interventions: Drug: Lacteol fort
- SLIT Group (Experimental): included 15 children who received SLIT for 6 months. Standardized Timothy Grass Pollen (Phleum pratense)
  Interventions: Drug: Standardized Timothy Grass Pollen
- Combined treatment Group (Experimental): included 15 children who received probiotics and SLIT. A drug called Lacteol fort was administered A sachet was taken once daily for 3 months . Standardized Timothy Grass Pollen was taken for 6 months
  Interventions: Drug: Lacteol fort and Standardized Timothy Grass Pollen

INTERVENTIONS:
Drug: Lacteol fort — Lacteol fort is a drug containing lactobacilli
  Arms: Probiotic Group
Drug: Standardized Timothy Grass Pollen — SLIT includes 2 phases build up and maintenance phases. (Jubilant HollisterStier LLC 14110 Collections Drive, Chicago USA) .
  Arms: SLIT Group
Drug: Lacteol fort and Standardized Timothy Grass Pollen — Lacteol fort is a drug containing lactobacilli and the Standardized Timothy Grass Pollen includes 2 phases build up and maintenance phases.
  Arms: Combined treatment Group

SUMMARY:
The investigators aimed to explore miRNA-155 change in response to sublingual immunotherapy (SLIT), probiotics and combined treatment with SLIT and probiotics in AR children.

DETAILED DESCRIPTION:
Allergic rhinitis (AR) is an inflammatory state characterized by a disturbance of immunoregulatory mechanisms that leads to an amplified T helper "Th-2" response. Micro-RNAs (miRNAs) are short single-stranded RNA molecules that post transcriptionally control gene expression and can mediate allergic process. The aim of this study was to explore miRNA-155 change in response to sublingual immunotherapy (SLIT), probiotics and combined treatment with SLIT and probiotics in AR children.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5-18 years
* Diagnosed as having AR
* With positive skin test to grass pollen

Exclusion Criteria:

* Anatomical abnormalities of upper respiratory tract,
* Previous immunotherapy,
* Clinically significant inﬂammatory diseases,
* Malignancies,
* Chronic treatment with systemic corticosteroids or immune suppressive drugs

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-03-10 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Total nasal symptom score between before and after treatment | 6 months
  Total Nasal Symptom Score was evaluated for the three groups at the start of the study and after 6 months. TNSS is the sum of scores for each of nasal obstruction, sneezing, nasal itching, and rhinorrhea at each time point, by means of a four-point scale (0-3) . TNSS is estimated by addition of the score for each of the symptoms to a total out of 12

SECONDARY OUTCOMES:
Serum miR-155 expression at the start and end of the study | 6 months
  Serum miR-155 expression was measured for the three groups by quantitative real time PCR

CONTACTS AND LOCATIONS:
Overall Officials: Randa Sedeek, Study Chair — Medical Microbiology and Immunology
Locations (1):
- Zagazig university, Zagazig, Sharqia Province, Egypt

REFERENCES:
- [Background] Livak KJ, Schmittgen TD. Analysis of relative gene expression data using real-time quantitative PCR and the 2(-Delta Delta C(T)) Method. Methods. 2001 Dec;25(4):402-8. doi: 10.1006/meth.2001.1262. PMID 11846609
- [Background] Cox L. Sublingual immunotherapy and allergic rhinitis. Curr Allergy Asthma Rep. 2008 Apr;8(2):102-10. doi: 10.1007/s11882-008-0019-5. PMID 18417051